CLINICAL TRIAL: NCT03835936
Title: Immediate Effects and Safety of High-frequency Chest Wall Oscillation Compared to Airway Clearance Techniques in Non-hospitalized Infants With Acute Viral Bronchiolitis
Brief Title: Treatment of Pediatric Bronchiolitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guadarrama Hospital (Other)
Collaborators: Fisiobronquial Clínicas (Other)
Responsible Party: Principal Investigator, J. Nicolas Cuenca Zaldivar, Rehabilitation Service Principal Investigator, Guadarrama Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5.0
Record Dates: First submitted 2019-02-07; First posted 2019-02-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Bronchiolitis
Keywords: Physical Therapy; Respiratory; Pediatric
MeSH Terms: conditions — Bronchiolitis

STUDY DESIGN:
Intervention Model Description: Single-blind controlled clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual maneuvers physiotherapy (Active Comparator): The protocol of physiotherapy treatment techniques consists of 20 minutes of FR based on prolonged slow expiration and cough provoked.
  Interventions: Other: Manual maneuvers physiotherapy group
- High frequency compression chest wall (Experimental): The protocol consists in the application of the Smart Vest® device for high frequency compression of the chest wall, with a fixed frequency of 13 Hz and a time of 15 minutes. Then during 20 minutes will apply the same protocol as in the manual maneuvers group.
  Interventions: Other: High frequency compression of the chest wall group; Other: Manual maneuvers physiotherapy group

INTERVENTIONS:
Other: High frequency compression of the chest wall group — The protocol in the high frequency compression of the chest wall group device consists of the Smart Vest® application, with a fixed frequency of 13 Hz and a time of 15 minutes. The selected mode will be the normal (fixed parameters) and the pressure of 4 units (12 cm H2O). The patient remains seated on his parents, and with a cotton garment between the vest and the skin of the patient to prevent skin lesions.
  Arms: High frequency compression chest wall
Other: Manual maneuvers physiotherapy group — 20 minutes of manual maneuvers physiotherapy based on prolonged slow expiration: passive technique of expiratory help applied to the baby through a slow thoracic-abdominal pressure that begins at the end of spontaneous expiration and continues to the residual volume. The physiotherapist through the cough provoked or stimulation of the trachea gets expectoration of sputum, to be able to assess its weight.

SUMMARY:
Bronchiolitis (BQ) is the acute viral infection of the tract respiratory syndrome in infants that affects the bronchioles of babies under 24 months of age. Respiratory physiotherapy (RF) appears as a treatment measure complementary in the clinical guidelines and consensus on the management of the BQ.

DETAILED DESCRIPTION:
Once each patient legal guardians has signed the informed consent document and it has been verified that the inclusion criteria are met, it will be assigned the same identification number (ID) that is related to its Clinical History (CH) by simple coding; custody of the file with the relationship of each ID with its CH will be the responsibility of the principal investigator.

The assignment will be made at the time of query according to a table of random numbers previously established and that it will only be known by physiotherapists.

Before starting the treatment protocol, a blind evaluator who does not know the treatment to which the patient is assigned, classifies the child according to the initial score of clinical severity proposed by Wang, in addition to the measurement of SO2 and frequency heart rate through a pulse oximeter. The measurement of the amount of sputum collected in a meter measuring cup, once the respiratory physiotherapy session is finished, it will be done in a calibrated weight in both groups.

The protocol in the manual maneuvers group consists of 20 minutes of FR based on prolonged slow expiration and coughing provoked. Is apassive technique of expiratory help applied to the baby through a slow thoracic-abdominal pressure that begins at the end of spontaneous expiration and continues to the residual volume. The physiotherapist through the cough provoked or stimulation of the trachea gets expectoration of sputum, to be able to assess its weight.

The protocol in the high frequency compression chest wall group consists of the same protocol as the respiratory physiotherapy Group plus high frequency compression chest wall applied with Smart Vest® device, with a fixed frequency of 13 Hz and a time 15 min. The selected mode will be the normal (fixed parameters) and the pressure of 4 units (12 cm H2O). The patient remains seated on his parents, and with a cotton garment between the vest and the skin of the patient to prevent skin lesions.

Attention must be paid during maneuvers to maintain a position of infant in supine decubitus in 30 degrees of slope, to avoid episodes of gastroesophageal reflux and decrease the risk of vomiting.

Criteria for cessation of physiotherapeutic intervention, alterations will be considered abrupt of the respiratory rhythm (brady or tachypnea), stare, ocular revulsion, hiccups or hypertonia and changes in skin color (pallor or cyanosis). In addition to these manifestations clinics, it is established that if the parent or legal guardian so requires, the the application of the protocol.

After 10 and 20 minutes of finishing both groups, the doctor again makes a measurement of mucus volume, SO2, heart and respiratory rate, and classify again according to the criteria of Wang's clinical severity scale.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet the following inclusion criteria:

* Have an age between 2 months and 12 months.
* Have a medical diagnosis of the first episode of BQ.
* Have the informed consent signed by the child's legal guardians.

Exclusion Criteria:

The criteria of exclusion are:

* BQ in acute phase with score> 9 according to Wang clinical scale.
* Associated cardiac, neurological or traumatic pathology.
* Previous hospitalization for wheezing.
* Medical diagnosis of recurrent sibilant.

Ages: 2 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-05-10 (Actual); Study Completion 2019-05-10 (Actual)

PRIMARY OUTCOMES:
Wang clinical severity scale | 12 weeks
  The clinical severity scale of Wang evaluates the respiratory rate, the presence of wheezing and intercostal retraction, and the patient's general condition, puncturing each dimension from 0 (the possible state) to 3 (values within normal), in addition to offer different cut points for children with more or less than 6 months.

SECONDARY OUTCOMES:
Oxygen saturation | 12 weeks
  Measured by a pulse oximeter (Radical 7 Touchscreen by Massimo®, Masimo Corporation, Irvine, CA).
Heart rate | 12 weeks
  Measured by a pulse oximeter (Radical 7 Touchscreen by Massimo®, Masimo Corporation, Irvine, CA).
Amount of sputum | 12 weeks
  The measurement of the amount of sputum collected in a metric measuring cup, once the session is finished, will be done in a calibrated weight

CONTACTS AND LOCATIONS:
Overall Officials: J. Nicolas Cuenca Zaldivar, Principal Investigator — Guadarrama Hospital
Locations (1):
- J.Nicolas Cuenca Zaldivar, Guadarrama, Madrid, Spain

REFERENCES:
- [Derived] Roque-Figuls M, Gine-Garriga M, Granados Rugeles C, Perrotta C, Vilaro J. Chest physiotherapy for acute bronchiolitis in paediatric patients between 0 and 24 months old. Cochrane Database Syst Rev. 2023 Apr 3;4(4):CD004873. doi: 10.1002/14651858.CD004873.pub6. PMID 37010196
- [Derived] Gonzalez-Bellido V, Velaz-Baza V, Blanco-Moncada E, Del Carmen Jimeno Esteo M, Cuenca-Zaldivar JN, Colombo-Marro A, Donadio MVF, Torres-Castro R. Immediate Effects and Safety of High-Frequency Chest Wall Compression Compared to Airway Clearance Techniques in Non-Hospitalized Infants With Acute Viral Bronchiolitis. Respir Care. 2021 Mar;66(3):425-433. doi: 10.4187/respcare.08177. Epub 2020 Nov 3. PMID 33144386